CLINICAL TRIAL: NCT01523912
Title: Ablation of Gastric Dysplastic Mucosa by a Novel Endoscopic Radiofrequency Device.
Brief Title: Radiofrequency Ablation for the Treatment of Gastric Dysplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Francisco Baldaque-Silva, Principal Investigator, Hospital Sao Joao
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gastric ablation; SG.HSJ.FMUP.01.2012 (Other: Hospital Sao Joao)
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Dysplasia; Neoplasia
Keywords: radiofrequency ablation; gastric dysplasia; gastric neoplasia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gastric RFA (Experimental): Ablation of gastric dysplastic mucosa
  Interventions: Device: Radiofrequency ablation of dysplastic mucosa (HALO)

INTERVENTIONS:
Device: Radiofrequency ablation of dysplastic mucosa (HALO) — Gastric ablation is performed using the HALO Ablation System (BÂRRX Medical Inc., Sunnyvale, CA, USA). A HALO90 ablation catheter, which is mounted on the tip of an endoscope, is used. Radiofrequency energy is delivered at 40 W/cm2 and 15 J/cm2 via a 13 x 20 mm electrode. All patients will have two RFA sessions 8 weeks apart with the same area being ablated in consecutive endoscopies. The precise area to ablated in the second RFA session is determined by referring to careful measurements that utilized gastric landmarks (a typical notation may specify that the lesion extends from 2 to 5 cm proximal of the pylorus in the 5 o'clock position and is 4 cm wide) as well as to digital image recordings that are taken during the first RFA.
  Other Names: Halo; RFA

SUMMARY:
The finding of gastric dysplasia not associated with macroscopic lesions (DNAML) or the follow-up of dysplasia after endoscopic resection (DAER) is a challenging dilemma. In the last few years, radiofrequency ablation (RFA) has become a recognized tool in the treatment of dysplastic Barrett's esophagus, but its use in gastric dysplasia has not yet been studied. The investigators aim to study the efficacy, safety and tolerability of RFA in the treatment of dysplastic gastric mucosa.

DETAILED DESCRIPTION:
Gastric cancer is the fourth most common cancer and the second leading cause of cancer related death worldwide. The 10-year survival of patients with this malignancy is 20% due to advanced disease at the time of diagnosis. Screening programs in countries with a high incidence of gastric neoplasia aim to detect early stage cancer, suitable for curative treatment. Well-differentiated dysplastic gastric lesions limited to the mucosa (when non-ulcerated or ulcerated and less than 3 cm) or limited to the superficial submucosa (when less than 3 cm and with no lymphatic or vascular invasion) have a negligible risk of lymph node metastasis and are suitable for endoscopic curative treatment.

Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) have been increasingly used in this setting with promising results. However, even with these advanced techniques, en bloc and R0 resection is not possible in up to 13-15% and 16-26% of the cases, respectively. The presence of dysplasia after endoscopic resection (DAER) in the post-resection scar presents a challenging dilemma due to the technical difficulty, and associated complications, of performing subsequent EMR/ESD in fibrotic tissue. Another issue of concern is the presence of gastric dysplasia not associated with macroscopic lesions (DNAML). In such cases, a targeted endoscopic treatment is difficult and clinical management is not standardized.

Radiofrequency ablation (RFA) has been increasingly advocated for the treatment of dysplastic Barrett's esophagus (BE) and early esophageal squamous cell carcinoma (ESCC), but its use in gastric dysplasia has not yet been tested. The investigators aim to study the role of gastric RFA in the treatment of DNAML and DAER.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of gastric dysplasia.
2. The lesion is no larger than 5 cm in diameter.
3. Age ≥ 18 years.
4. Subject is able to tolerate endoscopy and sedation.
5. Subject agrees to participate, fully understands content of the informed consent, and signs the informed consent form.

Exclusion Criteria:

1. Prior gastric irradiation or surgery.
2. Anti-platelet or anti-thrombotic medication use that can not be stopped for 7 days before and after RFA.
3. Gastric ulcers, fistulae, varices and malignancy.
4. History of alcohol and/or controlled substance dependency.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The % of patients with complete histological clearance of dysplasia. | 12 months

SECONDARY OUTCOMES:
Histological clearance of intestinal metaplasia | 12 months
Adverse event incidence | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Baldaque-Silva, MD, Principal Investigator — Hospital Sao Joao
Locations (1):
- Gastroenterology Department, Hospital de Sao Joao, Porto, Portugal